CLINICAL TRIAL: NCT02193581
Title: Non-invasive Melanoma Assessment Using a Topical Fluorescence Reagent and Optical Imaging: the MDS (Melanoma Detecting System)
Brief Title: Non-invasive Melanoma Assessment Using a Topical Fluorescence Reagent and Optical Imaging
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: OMS 001_HMO
Record Dates: First submitted 2014-07-08; First posted 2014-07-17 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Skin Lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspicious skin lesions.: Patients with a suspicious skin lesion referred for a biopsy are tested using MDS
  Interventions: Device: MDS

INTERVENTIONS:
Device: MDS — Patients with a suspicious lesion, referred for a biopsy is tested using MDS.

SUMMARY:
The use of MDS to access the presence of melanoma in the skin.

DETAILED DESCRIPTION:
A topical agent is applied to suspicious skin lesions and imaged. The images are analyzed to provide a score that correlates with the probability for the presence of melanoma in the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with skin lesion with one or more of the ABCDE features and recommended for a skin biopsy.
* The lesion is accessible to the imaging device, with at least 1 cm of skin around the lesion that is accessible to the MDS.
* Male and female ≥ 21 years old.
* Subject is capable of giving written informed consent.
* Primary excision.

Exclusion Criteria:

* The lesion is less than 1 cm from the eyes.
* The lesion is on the palms of hands or soles of the feet.
* Mucosal lesion.
* Pregnant females.
* Low study procedure compliance.
* Patients who are mentally or physically unable to comply with all aspects of the study.
* Undergoing chemotherapy.
* Minor or legally incompetent and not able to sign the consent form.
* Patient previously tested by MDS and was diagnosed with melanoma during the study.
* Sensitivity to fluorescein

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual referred by a dermatologist or plastic surgeon for a skin biopsy or lesion excision.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The MDS produces a score between 1 to 10. | 28 days
  The score is a composite of the images of the mole, plus demographic and clinical information. The score is ranked from 1 to 10, with 1 being the lowest risk for melanoma, and 10 being the highest risk.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Merims, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel